CLINICAL TRIAL: NCT02420912
Title: Nivolumab Combined With Ibrutinib for Relapsed, Refractory or High-Risk Untreated Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Nivolumab and Ibrutinib in Treating Patients With Relapsed, Refractory, or High-Risk Untreated Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Richter Transformation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0931; NCI-2015-00844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0931 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Loss of Chromosome 17p; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Richter Syndrome
MeSH Terms: conditions — Chromosome 17 deletion; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort I (nivolumab, ibrutinib) Chronic Lymphocytic Leukemia (CLL) (Experimental): Patients receive nivolumab IV over 1 hour on days 1 and 15 and ibrutinib PO QD on days 1-28 of courses 2-24. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort II (nivolumab, previous ibrutinib) Chronic Lymphocytic Leukemia (CLL) (Experimental): Patients receive nivolumab as in Cohort I and continue previous ibrutinib treatment.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort III (nivolumab, ibrutinib) Richters Transformation (RT) (Experimental): Patients receive nivolumab and ibrutinib as in cohort I. Ibrutinib may be given earlier than course 2 in case of worsening disease after discussion with study principal investigator. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab and ibrutinib work when given together in treating patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, or Richter transformation that has come back after a period of improvement (relapsed), does not respond to treatment (refractory), or is at high risk of spreading and has not been treated. Immunotherapy with monoclonal antibodies, such as niolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving nivolumab together with ibrutinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy (response rate) of nivolumab in combination with ibrutinib in patients with relapsed/refractory or high-risk untreated chronic lymphocytic leukemia (CLL).

II. Determine the response rate (complete response [CR]/complete response with incomplete marrow recovery [CRi]) by 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria. (Cohort I) III. Determine the conversion rate from partial response (PR) to CR/CRi by 2008 IWCLL criteria. (Cohort II) IV. Determine the response rate (CR/CRi). (Cohort III)

SECONDARY OBJECTIVES:

I. To determine the safety of nivolumab in combination with ibrutinib in patients with relapsed, refractory or high-risk untreated CLL/Richter transformation (RT).

II. To determine the progression-free survival of patients with relapsed, refractory or high-risk untreated CLL/RT treated with nivolumab in combination with ibrutinib.

III. To determine the overall survival of patients with relapsed, refractory or high-risk untreated CLL/RT treated with nivolumab in combination with ibrutinib.

EXPLORATORY OBJECTIVES:

I. To study immunological and molecular changes in peripheral blood, lymph node, and bone marrow in response to nivolumab and ibrutinib therapy.

OUTLINE: Patients are assigned to 1 of 3 treatment cohorts.

COHORT I (NO CURRENT IBRUTINIB TREATMENT): Patients receive nivolumab intravenously (IV) over 1 hour on days 1 and 15 and ibrutinib orally (PO) once daily (QD) on days 1-28 of courses 2-24. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

COHORT II (IBRUTINIB TREATMENT > 9 MONTHS): Patients receive nivolumab as in Cohort I and continue previous ibrutinib treatment.

COHORT III (RICHTER TRANSFORMATION): Patients receive nivolumab and ibrutinib as in cohort I. Ibrutinib may be given earlier than course 2 in case of worsening disease after discussion with study principal investigator. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity

* Note: After 3 cycles of treatment, nivolumab administration may be decreased to once every 4 weeks in all cohorts, in consultation with the study principal investigator.

After completion of study treatment, patients are followed up monthly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have a diagnosis of CLL or small lymphocytic lymphoma (SLL), refractory to or relapsed after at least one prior standard therapy or untreated with deletion (del)(17p) by fluorescence in-situ hybridization (FISH) (high-risk cytogenetics) and have an indication for treatment by IWCLL 2008 criteria (Cohort 1) OR have been on ibrutinib for at least 9 months with measurable persistent disease (absolute lymphocyte count [ALC] > 4 K/muL, any lymph node > 1.5 cm by computed tomography [CT] scan, or > 30% lymphocytes on bone marrow aspirate differential) (Cohort 2), OR patients will have a diagnosis of RT, refractory to and/or relapsed after at least one prior standard therapy or untreated with del(17p) by FISH (high-risk cytogenetics) (Cohort 3)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x upper limit of normal (ULN); for patients with Gilbert's disease, total bilirubin up to =< 3 x ULN is allowed provided normal direct bilirubin
* Serum creatinine =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception method during the study and for 23 weeks following the last dose of the study drugs; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy; males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drugs
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years; patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses); if patients have another malignancy that was treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center and after consultation with the principal investigator
* Any major surgery, radiotherapy, cytotoxic chemotherapy, biologic therapy, immunotherapy, immunomodulatory drugs, experimental therapy within 4 weeks prior to the first dose of the study drugs; Note: prior therapy with anti cluster of differentiation (CD)20 monoclonal antibody, anti CD52 monoclonal antibody, and lenalidomide are allowed; for oral targeted therapies (such as idelalisib, venetoclax), a washout of 3 days is allowed
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 2 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association functional classification
* History of stroke or cerebral hemorrhage within 2 month
* Patients who have uncontrolled hypertension (defined as sustained systolic blood pressure >= 160 mmHg or diastolic >= 100 mmHg)
* Known evidence of active cerebral/meningeal CLL; patients may have history of central nervous system (CNS) leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of registration
* Active, uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring steroid therapy
* Patients with autoimmune diseases are excluded: patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus, Wegener's granulomatosis)
* Patients with previous allogeneic stem cell transplant (SCT) within 6 months or with active acute or chronic graft-versus host disease are excluded; patients must be off immunosuppression for graft-versus host disease (GVHD) for at least 30 days before cycle 1 day 1
* Patients with organ allografts (such as renal transplant) are excluded
* History of interstitial lung disease or pneumonitis
* Patients who are on high dose steroid (> 10 mg daily of prednisone or equivalent) or immune suppression medications; Note: patients on high-dose steroids (doses > 10mg/day of prednisone or equivalent) or immune suppression medications are eligible provided these drugs are discontinued at least 3 days prior to starting on the study drugs
* Patients with uncontrolled active infection (viral, bacterial, and fungal) are not eligible
* Current or chronic hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Patient is pregnant or breast-feeding
* Concurrent use of investigational therapeutic agent
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) family 3, subfamily A (3A) inhibitor
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain N, Senapati J, Thakral B, Ferrajoli A, Thompson P, Burger J, Basu S, Kadia T, Daver N, Borthakur G, Konopleva M, Pemmaraju N, Parry E, Wu CJ, Khoury J, Bueso-Ramos C, Garg N, Wang X, Lopez W, Ayala A, O'Brien S, Kantarjian H, Keating M, Allison J, Sharma P, Wierda W. A phase 2 study of nivolumab combined with ibrutinib in patients with diffuse large B-cell Richter transformation of CLL. Blood Adv. 2023 May 23;7(10):1958-1966. doi: 10.1182/bloodadvances.2022008790. PMID 36287248
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
Started | 7 | 3 | 26
Completed | 7 | 3 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT) | Total
Number analyzed (Participants) | 7 | 3 | 26 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 14 | 22
  >=65 years | 2 | 0 | 12 | 14
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 70] | 64 [55 to 65] | 65 [47 to 88] | 64 [42 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 11 | 13
  Male | 5 | 3 | 15 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 5 | 3 | 21 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 26 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response for Cohorts 1 and 3
Description: Response is Complete Response (CR) + Partial Response (PR). CR = Peripheral blood Lymphocytes <4000/uL, no lymphadenopathy, no hepatomegaly or splenomegaly by exam or scan, absence of symptoms, neutrophils > 1,500/uL, Platelets > 1000,000/uL, hemoglobin > 11.0 g/dl (untransfused) and normocellular bone marrow < 30% nucleated cells being lymphocytes, no lymphoid nodules. PR = 1 for >/= 2 months: >/= 50% decrease in peripheral lymphocyte count from baseline, >/= 50% reduction in lymphadenopathy, >/= 50% reduction in pretreatment enlargement of the spleen or liver by scan. Additionally for PR must have 1 of the following for >/= 2 months: Neutrophils > 1,500/uL, Platelets > 100,000/uL or >/= 50% improvement over baseline or Hemoglobin > 11.0 g/dl (untransfused) or >/= 50% improvement over baseline. Additionally if patients fufill CR but have one of the following, be considered a PR: bone marrow nodules or persistent anemia, thrombocytopenia, neutropenia unrelated to disease.
Time Frame: Up to 12 months
Population: This outcome measure was only designed for those participants in cohort 1 and 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
Number analyzed (Participants) | 7 | 0 | 26
Participants | 5 |  | 10

2. Primary Outcome: Number of Participants in Cohort 2 to Convert From a Partial Response (PR) to Complete Response (CR)
Description: Complete Response (CR) = Peripheral blood Lymphocytes <4000/uL, no lymphadenopathy, no hepatomegaly or splenomegaly by exam or scan, absence of symptoms, neutrophils > 1,500/uL, Platelets > 1000,000/uL, hemoglobin > 11.0 g/dl (untransfused) and normocellular bone marrow < 30% nucleated cells being lymphocytes, no lymphoid nodules. Partial Response (PR) = 1 for >/= 2 months: >/= 50% decrease in peripheral lymphocyte count from baseline, >/= 50% reduction in lymphadenopathy, >/= 50% reduction in pretreatment enlargement of the spleen or liver by scan. Additionally for PR must have 1 of the following for >/= 2 months: Neutrophils > 1,500/uL, Platelets > 100,000/uL or >/= 50% improvement over baseline or Hemoglobin > 11.0 g/dl (untransfused) or >/= 50% improvement over baseline. Additionally if patients fufill CR but have one of the following, be considered a PR: bone marrow nodules or persistent anemia, thrombocytopenia, neutropenia unrelated to disease.
Time Frame: Up to 12 months
Population: This outcome measure was designed for participants from Cohort 2, already on ibrutinib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
Number analyzed (Participants) | 0 | 3 | 0
Participants |  | 1 |

3. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start until date of death due to any cause or last Follow-up. Survival will be presented by median survival, which is the time point at which the cumulative survival drops below 50%. If there is no median survival (not reached), it means the cumulative survival was more than 50%.
Time Frame: Up to 6 years, 7 months
Population: Two participants in Cohort 3 were not evaluable for response.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
Number analyzed (Participants) | 7 | 3 | 24
months | NA [8.2 to 79.0] — The median overall survival for Cohort 1 was Not Reached. insufficient number of participants with events | NA [78.0 to 79.0] — The median overall survival for Cohort 2 was Not Reached. insufficient number of participants with events and zero patients died while they were onstudy. | NA [1 to 19] — The median overall survival for Cohort 3 was Not Reached. insufficient number of participants with events

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 6 years, 7 months
Population: Two participants in Cohort 3 were not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
Number analyzed (Participants) | 7 | 3 | 24
Months | 50.1 [4.6 to 79.0] | 22.3 [7.8 to 46.7] | 15 [3.5 to 17.5]

ADVERSE EVENTS:
Time Frame: Up to 6 years, 7 months
Arm/Group | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT)
All-Cause Mortality (participants affected / at risk) | 3/7 | 0/3 | 13/26
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/3 | 15/26
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 19/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) (N=7) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) (N=3) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT) (N=26)
Abdominal pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (8)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Nivolumab, Ibrutinib) Chronic Lymphocytic Leukemia (CLL) (N=7) | Cohort II (Nivolumab, Previous Ibrutinib) Chronic Lymphocytic Leukemia (CLL) (N=3) | Cohort III (Nivolumab, Ibrutinib) Richters Transformation (RT) (N=26)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acute Otitis Media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 4 (6) | 0 (0) | 6 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4)
Decreased Hearing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 5 (6)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 3 (7)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Nervous system disorders (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (5) | 3 (4) | 4 (7)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 8 (8)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2) | 3 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sweats (General disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0) | 2 (3)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Weight loss (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT02420912/Prot_SAP_000.pdf